CLINICAL TRIAL: NCT01659307
Title: The Effect of Aspirin on REducing iNflammation in Human in Vivo Model of Acute Lung Injury
Acronym: ARENA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: The Intensive Care Society United Kingdom (Unknown); Northern Ireland Clinical Trials Unit (Other); Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Professor Danny McAuley, Professor of Intensive care Medicine, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11127DMcA-AS; 2012-001589-13 (EudraCT Number)
Record Dates: First submitted 2012-08-04; First posted 2012-08-07 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Acute Lung Injury
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Aspirin
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aspirin 75mg (Active Comparator): Aspirin 75mg once daily for 7 days. Administered by mouth.
  Interventions: Drug: Aspirin 75mg
- Aspirin 1200mg (Active Comparator): Asprin 600mg twice daily for 7 days. Administered by mouth.
  Interventions: Drug: Aspirin 1200mg
- Lactose powder (Placebo Comparator): Placebo for 7 days. Administered by mouth.
  Interventions: Drug: Lactose powder

INTERVENTIONS:
Drug: Aspirin 75mg — Subjects randomised to aspirin 75mg will receive 1 container containing aspirin 75mg and 1 container containing placebo for the morning and 2 containers containing placebo for the evening. Subjects will take one capsule from each container in the morning and one capsule from each container in the evening.
  Arms: Aspirin 75mg
Drug: Lactose powder — Subjects randomised to placebo will receive 4 containers of placebo, 2 containers containing placebo for the morning and 2 containers containing placebo for the evening. Subjects will take one capsule from each container in the morning and one capsule from each container in the evening.
  Arms: Lactose powder
Drug: Aspirin 1200mg — Subjects randomised to aspirin 600mg 12 hourly will receive 2 containers of aspirin 300mg each for the morning and 2 containers of aspirin 300mg each for the evening. Subjects will take one capsule from each container in the morning and one capsule from each container in the evening.
  Arms: Aspirin 1200mg

SUMMARY:
This is a double-blind, placebo-controled, randomized trial to investigate if aspirin pre-treatment has anti-inflammatory effects in a model of acute lung injury induced by inhaled endotoxin (LPS) in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Age < 18 years
* Pregnancy or breast feeding or woman of childbearing potential not using
* adequate contraception.
* Participation in a clinical trial of an investigational medicinal product within 30 days
* Consent declined Aspirin or non steroidal anti-inflammatory (NSAID) use in the past 4 weeks
* History of asthma
* Known aspirin or NSAID hypersensitivity
* History of peptic ulcer disease
* Platelet count < 150 x 106/ml
* Aspirin resistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2012-09; Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Bronchoalveolar lavage IL-8 concentration | 6 hrs after LPS inhalation

SECONDARY OUTCOMES:
Alveolar inflammatory response biomarkers | 6 hrs after LPS inhalation
Plasma inflammatory response biomarkers | 6 and 24 hrs after LPS inhalation
Alveolar epithelial and endothelial function and injury biomarkers | 6 hrs after LPS inhalation
Lipid inflammatory mediators | 6 and 24 hrs after LPS inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Danny McAuley, Principal Investigator — Queens University, Belfast
Locations (1):
- Belfast Health and Social Care Trust, Belfast, United Kingdom

REFERENCES:
- [Derived] Hamid U, Krasnodembskaya A, Fitzgerald M, Shyamsundar M, Kissenpfennig A, Scott C, Lefrancais E, Looney MR, Verghis R, Scott J, Simpson AJ, McNamee J, McAuley DF, O'Kane CM. Aspirin reduces lipopolysaccharide-induced pulmonary inflammation in human models of ARDS. Thorax. 2017 Nov;72(11):971-980. doi: 10.1136/thoraxjnl-2016-208571. Epub 2017 Jan 12. PMID 28082531
- [Derived] Toner P, McAuley DF, Shyamsundar M. Aspirin as a potential treatment in sepsis or acute respiratory distress syndrome. Crit Care. 2015 Oct 23;19:374. doi: 10.1186/s13054-015-1091-6. PMID 26494395
- [Derived] Curley GF, McAuley DF. Stem cells for respiratory failure. Curr Opin Crit Care. 2015 Feb;21(1):42-9. doi: 10.1097/MCC.0000000000000171. PMID 25486575